CLINICAL TRIAL: NCT04224571
Title: Chinese Children Cancer Group Relapsed Acute Lymphoblastic Leukemia 2017 Study
Brief Title: CCCG Relapsed Acute Lymphoblastic Leukemia 2017 Study in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Shanghai Children's Medical Center (Other)
Responsible Party: Principal Investigator, Prof. LI Chi Kong, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKCH-REC-2019-006
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse
Keywords: Relapsed ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bortezomib; Rituximab

STUDY DESIGN:
Intervention Model Description: Prospective and Non-randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rituximab and bortezomib (Experimental): to test whether adding rituximab in CD20 positive patients will have improvement in remission rate. (this arm terminated in October 2020) to add bortezomib in high risk patients at Induction to improve remission rate.
  Interventions: Drug: Bortezomib Injection; Drug: rituximab injection

INTERVENTIONS:
Drug: Bortezomib Injection — Bortezomib: patients with BM relapsed, add for 4 doses on D1,4,7, 11 in induction; dosage 1.3 mg/m2/dose as per parenteral;
  Other Names: Velcade
Drug: rituximab injection — Add rituximab in patients with CD20 positive ALL, rituximab: 6 doses of on D8,11of induction, D1,15 of consolidation1 and 2 with dosage 375 mg/m2 as parenteral (Terminated in Oct 2020)
  Other Names: Mab Thera

SUMMARY:
Relapsed acute lymphoblastic leukaemia (ALL) has a poorer outcome than newly diagnosed ALL patients with only about 40% overall survival after re-treatment. The study CCCG Relapsed ALL 2017 study will adopt the UK R3 study stratification and treatment backbone with two new agents added. There will be a 4-week induction, followed by two consolidation courses. High-risk patients will receive allogeneic stem cell transplant. While intermediate and standard risk groups will continue maintenance treatment for another 2 years or one year. New agents will be added aiming at improving survival outcome.

1. Study of adding anti-CD20 antibody (rituximab) with chemotherapy: CD20 is found to be expressed in 40-50% of B-lineage ALL, and rituximab has been studied in adult ALL with superior survival (75% vs 47%,). There is little experience of using rituximab in pediatric ALL thus a CCCG Relapsed ALL 2017 Study will perform the study assessing the remission rate and MRD response of CD20+ ALL treated with rituximab. Six doses of rituximab and will be monitored the week 5 MRD and relapse rate as study outcome.

   (This arm was terminated in October 2020 after interim analysis showing lack of efficacy)
2. Adding bortezomid during the induction: The very early or early bone marrow relapse has low remission rate. Previous case studies showed that Bortezomib, a proteasome inhibitor, may achieve remission in refractory ALL, 80% remission in B-ALL with combination of chemotherapy and bortezomib. Thus adding bortezomib, may improve the remission rate, thus bridging to allogeneic stem cell transplant. Adding bortezomib in the relapsed chemotherapy protocol may increase the toxicity and even treatment related mortality. In this protocol, we suggested to add during the induction therapy.

DETAILED DESCRIPTION:
Acute Lymphoblastic Leukemia (ALL) is now having over 80% event-free survival after frontline chemotherapy treatment. There is still 15-20% of patients having a relapse after initial control. Relapsed ALL is associated with lower second remission rate and also high chance of further relapse. Currently there are only a few large scale studies targeting this challenging disease. BFM Relapsed ALL studies have been organized since 1990s and have identified several important prognostic factors, including timing and site of relapse and also immunophenotyping. COG has performed several studies on relapsed ALL (AALL02P2, AALL0433, ADVL04P2) but the results are rather fragmented. Recently UK group conducted a nationwide randomized study, ALL R3 study, testing the type of anthracycline and prognostic value of minimal residual disease after induction therapy.

T-ALL relapse is having poor prognosis except for the late isolated extramedullary relapse. Long-term survival of T-ALL bone marrow relapse treated with chemotherapy is less than 10%, thus allogeneic stem cell transplant is always indicated. Whereas B-ALL has been better studied and the risk stratification of relapsed ALL is better defined.

According to previous studies, patients can be stratified into Standard, Intermediate and High-Risk groups based on site of relapse, time of relapse from first diagnosis and immunophenotyping. Early bone marrow relapse at less than 18-36 months from diagnosis is having the worst prognosis and is classified as HR. Those with late relapse at >36 months from diagnosis is in general having a better prognosis. Bone marrow relapse is having a poorer outcome as compared to isolated extramedullary relapse (IEM). Somehow combined marrow and extramedullary relapse appear to have a better prognosis than isolated bone marrow relapse. Early B-ALL marrow relapse was only having 15-30% long-term survival, and early B-ALL IEM around 30-50% survival.

Late B-ALL marrow relapse has a higher second remission rate of around 95% and also better long term survival of 50-60%. Late B-ALL IEM is having a better prognosis of up to 70-80% survival. Based on the above criteria, several study groups including BFM, UK and COG also adopted similar strategies of stratifying patients and delivered risk-adapted treatment, with some minor variation among these groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age at relapse less than 21 years and the age at initial diagnosis of ALL of Pre-B or T-lineage less than 18 years.
2. Confirmed diagnosis of relapse of leukemia according to definition as below:

Definitions of Relapse

* RELAPSE: Any recurrence of disease whether in marrow or extramedullary.
* (1) ISOLATED Bone Marrow Relapse: Patients with an M3 marrow (>25% blast) at any point after achieving remission without involvement of the CNS and/or testicles and/or other extramedullary sites. Relapsed should be confirmed by morphology, flow cytometry, FISH and/or cytogenetics. M2 marrow should have a repeat of bone marrow in 1-2 weeks to confirm M3 status unless the original cytogenetic clone reappears.

  (2) CNS Relapse: Positive cytomorphology and WBC ≥ 5/μL OR clinical signs of CNS leukemia such as facial nerve palsy, brain/eye involvement, or hypothalamic syndrome that are compatible with recurrent CNS leukemia than to alternative causes (e.g., viral infection with facial nerve palsy or chemotherapy toxicity). If any CSF evaluation shows positive cytomorphology and WBC < 5/μL, a second CSF evaluation is recommended within 2 - 4 weeks. While identification of a leukemic clone in CSF by flow cytometry (TdT, CD19, CD10, etc.) or FISH for diagnostic karyotypic abnormality may be useful, definitive evidence of CNS involvement (i.e. WBC ≥ 5/μL OR clinical signs of CNS leukemia) is required for the diagnosis of a CNS relapse.

  (3) TESTICULAR Relapse: Must be documented by testicular biopsy, if not associated with a marrow relapse.

  (4) ISOLATED Extramedullary (IEM) relapse: CNS and/or testicular relapse and/or other extramedullary sites such as skin with an M1 marrow. The presence of MRD in the bone marrow does NOT exclude IEM.

  (5) COMBINED Relapse: M2 or M3 marrow at any time after achieving remission with concomitant CNS and/or testicular relapse.

CNS Status:

CNS 1: In cerebral spinal fluid (CSF), absence of blasts on cytospin preparation, regardless of the number of white blood cells (WBCs).

CNS 2: In CSF, presence < 5/μL WBCs and cytospin positive for blasts, or ≥ 5/μL WBCs but negative by Steinherz/Bleyer algorithm:

CNS 2a: < 10/μL RBCs; < 5/μL WBCs and cytospin positive for blasts; CNS 2b: ≥ 10/μL RBCs; < 5/μL WBCs and cytospin positive for blasts; and CNS 2c: ≥ 10/μL RBCs; ≥ 5/μL WBCs and cytospin positive for blasts but negative by Steinherz/Bleyer algorithm (see below).

CNS3: In CSF, presence of ≥ 5/μL WBCs and cytospin positive for blasts and/or clinical signs of CNS leukemia:

CNS 3a: < 10/μL RBCs; ≥ 5/μL WBCs and cytospin positive for blasts; CNS 3b: ≥ 10/μL RBCs, ≥ 5/μL WBCs and positive by Steinherz/Bleyer algorithm (see below); CNS 3c: Clinical signs of CNS leukemia (such as facial nerve palsy, brain/eye involvement or hypothalamic syndrome).

Method of Evaluating Initial Traumatic Lumbar Punctures:

If the patient has leukemic cells in the peripheral blood and the lumbar puncture is traumatic and contains ≥ 5 WBC/μL and blasts, the following algorithm should be used to distinguish between CNS 2 and CNS 3 disease: CSF WBC > 2X Blood WBC CSF RBC Blood RBC

Exclusion Criteria:

1. Mature B ALL,
2. Poor Karnosky score

Ages: 3 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 208 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
remission rate | week 5 MRD and relapse rate
  bone marrow blast count < 5% and MRD <0.01%

SECONDARY OUTCOMES:
event-free survival rates | 2-year
  survive without relapse or death or second cancer, with or without HSCT
overall survival | 5 years
  survive without death event

CONTACTS AND LOCATIONS:
Overall Officials: Chi Kong LI, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pui CH, Carroll WL, Meshinchi S, Arceci RJ. Biology, risk stratification, and therapy of pediatric acute leukemias: an update. J Clin Oncol. 2011 Feb 10;29(5):551-65. doi: 10.1200/JCO.2010.30.7405. Epub 2011 Jan 10. PMID 21220611
- [Background] Tallen G, Ratei R, Mann G, Kaspers G, Niggli F, Karachunsky A, Ebell W, Escherich G, Schrappe M, Klingebiel T, Fengler R, Henze G, von Stackelberg A. Long-term outcome in children with relapsed acute lymphoblastic leukemia after time-point and site-of-relapse stratification and intensified short-course multidrug chemotherapy: results of trial ALL-REZ BFM 90. J Clin Oncol. 2010 May 10;28(14):2339-47. doi: 10.1200/JCO.2009.25.1983. Epub 2010 Apr 12. PMID 20385996
- [Background] Parker C, Waters R, Leighton C, Hancock J, Sutton R, Moorman AV, Ancliff P, Morgan M, Masurekar A, Goulden N, Green N, Revesz T, Darbyshire P, Love S, Saha V. Effect of mitoxantrone on outcome of children with first relapse of acute lymphoblastic leukaemia (ALL R3): an open-label randomised trial. Lancet. 2010 Dec 11;376(9757):2009-17. doi: 10.1016/S0140-6736(10)62002-8. Epub 2010 Dec 3. PMID 21131038
- [Background] Bertaina A, Vinti L, Strocchio L, Gaspari S, Caruso R, Algeri M, Coletti V, Gurnari C, Romano M, Cefalo MG, Girardi K, Trevisan V, Bertaina V, Merli P, Locatelli F. The combination of bortezomib with chemotherapy to treat relapsed/refractory acute lymphoblastic leukaemia of childhood. Br J Haematol. 2017 Feb;176(4):629-636. doi: 10.1111/bjh.14505. Epub 2017 Jan 24. PMID 28116786
- [Background] Maury S, Chevret S, Thomas X, Heim D, Leguay T, Huguet F, Chevallier P, Hunault M, Boissel N, Escoffre-Barbe M, Hess U, Vey N, Pignon JM, Braun T, Marolleau JP, Cahn JY, Chalandon Y, Lheritier V, Beldjord K, Bene MC, Ifrah N, Dombret H; for GRAALL. Rituximab in B-Lineage Adult Acute Lymphoblastic Leukemia. N Engl J Med. 2016 Sep 15;375(11):1044-53. doi: 10.1056/NEJMoa1605085. PMID 27626518
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074